NCT05216510 Document Date: 27July2022

# Statistical Analysis Plan

| Sponsor | Tonix Pharmaceuticals, Inc. |
|---|---|
| Protocol Title: | A Dose Finding Study for the Assessment of Delayed-type Hypersensitivity Reactions to SARS-CoV-2 Peptide Antigens in Uninfected Healthy Subjects, COVID-19 Convalescent Subjects, and COVID-19 Vaccinated Subjects "COVID-19 DTH" |
| Protocol Number: | TNX-CA-C201 |
| Document Version: | 1 |

# Approvals



Note: The date of the analysis plan is the date of the final approval signature.

Version 1 

# **Document Revision History**

| Revision History | | | |
|---|---|---|---|
| SAP Version # | Modification | Description and<br>Rationale | Superseded SAP<br>Version # |
| 1.0 | N/A | N/A | N/A |

Version 1 

# **Table of Contents**

| Ap | provals | | 1 |
|---|---|---|---|
| Do | cument | Revision History | 2 |
| Ta | ble of C | Contents | 3 |
| Lis | st of Ab | breviations | 5 |
| 1. | . Overview | | |
| 2. Study Objectives and Endpoints | | | |
| | 2.1. | Study Objectives | 7 |
| | 2.1.1. | Primary Objective | 7 |
| | 2.1.2. | Secondary Objectives | 7 |
| | 2.2. | Study Endpoints | 8 |
| | 2.2.1. | Efficacy Endpoints | 8 |
| | 2.2.2. | Safety Endpoints | 8 |
| | 2.3. | Modified Evaluation | 9 |
| 3. Overall Study Design and Plan | | rerall Study Design and Plan | 9 |
| | 3.1. | Overall Design | 9 |
| | 3.2. | Sample Size and Power | 10 |
| | 3.3. | Study Population | 10 |
| | 3.4. | Treatments Administered | 10 |
| | 3.5. | Method of Assigning Subjects to Treatment Groups | 10 |
| | 3.6. | Blinding and Unblinding. | 10 |
| | 3.7. | Schedule of Events | 10 |
| 4. | Sta | itistical Analysis and Reporting | 11 |
| | 4.1. | Introduction | 11 |
| 5. | Stı | udy Halting and Stopping Rules | 11 |
| 6. | An | alysis Populations | 11 |
| 7. | Ge | neral Issues for Statistical Analysis | 12 |
| | 7.1. | Statistical Definitions and Algorithms | 12 |
| | 7.1.1. | Baseline | 12 |
| | 7.1.2. | Adjustments for Covariates | 12 |
| | | Multiple Comparisons | 12 |
| | 7.1.4. | Handling of Dropouts or Missing Data | 12 |
| | 7.1.5. | Analysis Visit Windows | 12 |
| | 7.1.6. | Derived Variables | 12 |
| | | Data Adjustments/Handling/Conventions | |
| 8. | | ady Patients/Subjects and Demographics | |
| | 8.1. | Disposition of Patients/Subjects | |
| | 8.2. | Protocol Violations and Deviations | 14 |



# List of Abbreviations

| Abbreviation | Definition |
|---|---|
| AE | Adverse event |
| AESI | Adverse event of special interest |
| BMI | Body mass index |
| CANDIN® | Candida albicans skin test antigen for cellular hypersensitivity |
| COVID-19 | Coronavirus disease 2019 |
| CRF | Case report form |
| DTH | Delayed-type hypersensitivity |
| ELISpot | Enzyme-linked immune absorbent spot |
| FDA | Food and Drug Administration |
| GCP | Good clinical practices |
| GLP | Good laboratory practices |
| ICF | Informed consent |
| ICH | International Council for Harmonisation |
| ICS | Intracellural cytokine staining |
| IP | Investigational product |
| IRB | Institutional review board |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NP | Nasopharyngeal |
| PBMC | Peripheral blood mononuclear cells |
| PI | Principal investigator |

Version 1 

| Abbreviation | Definition |
|--------------|-------------------------------------------------|
| POC | Proof-of-Concept |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SOC | System Organ Class |
| SAS | Statistical Analysis System |
| SARS-CoV-2 | Severe acute respiratory syndrome coronavirus 2 |
| Th | T helper cell |
| TEAE | Treatment-emergent adverse event |
| WHO | World Health Organization |

Version 1 

#### 1. Overview

This statistical analysis plan (SAP) describes the planned analysis and reporting for Tonix Pharmaceuticals, Inc. protocol number TNX-CA-C201 (A Dose Finding Study for the Assessment of Delayed-type Hypersensitivity Reactions to SARS-CoV-2 Peptide Antigens in Uninfected Healthy Subjects, COVID-19 Convalescent Subjects, and COVID-19 Vaccinated Subjects "COVID-19 DTH"), dated 07-Dec-2021, version Final v2.0, amendment 01. Reference materials for this statistical plan include the protocol and the accompanying sample data collection documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials (ICH, 1998). All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association (ASA, 2018) and the Royal Statistical Society (RSS, 2014), for statistical practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc or unplanned, exploratory analysis performed will be clearly identified as such in the final CSR.

The final clinical database cannot be locked until the final SAP has been approved and signed.

## 2. Study Objectives and Endpoints

#### 2.1. Study Objectives

## 2.1.1. Primary Objective

The main objectives of the study are to evaluate the safety of intradermally-injected synthesized TNX-2100 SARS-Co V-2 peptide antigens and to assess the presence of DTH reactions in response to intradermal injection of synthesized TNX-2100 SARS-Co V-2 peptide antigens.

## 2.1.2. Secondary Objectives

The secondary objectives are:

- To estimate sensitivity and specificity of test as a marker of active or recovered infection relative to clinical history of infection.
- To identify the optimal synthesized SARS-CoV-2 peptide antigens and concentration for sensitive and specific DTH reaction.
- To identify the optimal timepoint for assessment of the DTH reaction.

Version 1 

• To correlate the DTH reaction with the adaptive T-cell immune response to SARS-CoV-2.

# 2.2. Study Endpoints

## 2.2.1. Efficacy Endpoints

### 2.2.1.1. Primary Efficacy Endpoint

The primary efficacy endpoint of this study is the maximal area of induration ≥5 mm at injection sites on the volar aspect of the forearms at 48 hours, 72 hours, and 96 hours post skin test administration.

### 2.2.1.2. Secondary Efficacy Endpoints

The secondary efficacy endpoints of this study include the following:

- Correlation of DTH reaction to clinical history of prior SARS-CoV-2 infection.
- Correlation of DTH reaction to adaptive T-cell immune response to SARS-CoV-2 assessed by T-Detect COVID Test (Adaptive Biotechnologies).
- Correlation of DTH reaction with in vitro assays of immune response including SARS CoV-2 antibody levels.
- Characterization of Th1 and Th2 responses by measuring cytokine production and cell surface T-cell phenotype markers by intracellular cytokine staining.

## 2.2.1.3. Exploratory Efficacy Endpoint

The exploratory efficacy endpoint is a characterization of Th17 response by enzyme linked immune assay.

#### 2.2.2. Safety Endpoints

Safety of intradermally administered TNX-2100 SARS-CoV-2 peptides, as measured by:

- Incidence of AEs.
  - O Clinically abnormal symptoms and other AEs will be assessed as defined in the FDA Guidance for Industry: "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" using a 4-point system (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, and Grade 4 = potentially life threatening).
  - Adverse events of systemic allergic reaction will be graded according to the World Allergy Organization Grading Scale for Systemic Allergic Reactions.
  - Local skin reactions will be captured by a subject self-reported 7-point Likert scales indicating severity of: erythema, pain, pruritis, and swelling.

Version 1 

- Protocol-defined adverse events of special interest (AESI):
  - o Anaphylactic reaction.
  - Enhanced disease from repeated exposure to SAR-CoV-2 (in subjects who have recovered from SARS-CoV-2 infection or in subjects recently vaccinated against SARS-CoV-2).

#### 2.3. Modified Evaluation

Because the outcome of area of induration for the DTH reactions was not as anticipated, the DTH reactions will not be statistically analyzed. Any primary, secondary, or exploratory efficacy endpoint will be omitted from the analysis and only safety will be assessed.

## 3. Overall Study Design and Plan

## 3.1. Overall Design

This will be a proof-of-concept (POC), dose finding, multi-cohort study designed to evaluate the safety of intradermally-injected synthesized TNX-2100 SARS-CoV-2 peptide antigens and assess the presence of DTH reactions in response to intradermal injection of synthesized TNX-2100 SARS-CoV-2 peptide antigens. This study will be conducted in a total of approximately 90 subjects (30 subjects per cohort) who are either uninfected/unexposed healthy individuals (Cohort 1), who are confirmed to have recovered from SARS-CoV-2 infection, independent of vaccination status (Cohort 2) or who have received a complete SARS-CoV-2 vaccine course with no known history of natural infection (Cohort 3).

The study will consist of a baseline/skin test administration at Visit 1 (Day 1) at which time baseline assessments are to be completed, the skin test is performed, and appropriate test samples are collected. Follow-up visits to monitor safety and evaluate the presence or absence of DTH reactions will be conducted per the following schedule: Visit 2 (Day 2); Visit 3 (Day 3); Visit 4 (Day 4); Visit 5 (Day 5). Safety monitoring will continue at Visit 6 (Day 30) and Visit 7 (Day 180) by telephone calls. The estimated study duration will be approximately 6 months. Photography of the injection site (volar forearms) after IP administration at Visit 1 and at Visit 3, 4, and 5, or unscheduled in person visits, will be used for safety documentation of local skin reaction, such as redness and swelling, or unexpected findings such as rash, blistering and necrosis, which require assessment by the designated Investigator.

Eligible subjects who provide written informed consent and who satisfy eligibility criteria will undergo a nasopharyngeal swab for a polymerase chain reaction (PCR) (reverse transcriptase [RT]-PCR or other) test to detect active SARS-CoV-2 infection. A laboratory PCR test or a sponsor approved rapid PCR test (such as the Accula<sup>TM</sup> RT-PCR test) may be used. If a laboratory PCR test is used, subjects will complete a Screening Visit between Day -2 and Day -1 to allow processing of the sample prior to the Baseline/Skin Test Administration Visit 1 (Day 1). The rapid PCR test can be performed at Visit 1 (Day 1) and is preferred to facilitate enrollment by reducing the number of required site visits. If the test result is negative, the subject will

Version 1 

proceed with the required blood draws followed by intradermal injection of the investigational products (IPs) and controls.

## 3.2. Sample Size and Power

Formal sample size calculations were not performed. The number of subjects were chosen based on feasibility and are considered sufficient to meet the study objectives. Approximately 90 subjects (30 subjects per cohort) will be enrolled.

## 3.3. Study Population

The study population consists of male and female adults, aged 18 to 65 years of age, inclusive. Subjects will be uninfected/unexposed healthy individuals (cohort 1), SARS-CoV-2 convalescent subjects (cohort 2), or SARS-CoV-2 vaccinated subjects (cohort 3).

## 3.4. Treatments Administered

Intradermal injections will be administered in two stages. At Stage 1, each subject will receive the diluent (negative control), followed by the "1:10 dilution" strength of TNX-2110, TNX 2120 and TNX 2130 in their left forearm, and a CANDIN® (positive control) in their right forearm. If no systemic adverse reactions or unusual local site reactions per the Principal Investigator's (PI) judgement are observed during 60 minutes after Stage 1 administration, the subjects will proceed to Stage 2.

At Stage 2, Subjects will receive the "undiluted" dose strength of TNX-2110, TNX-2120, TNX-2130 in the right forearm in the order and at the specific location. If no evidence of systemic adverse reactions or unusual local site reactions, per the PI's judgement, have occurred during the 30 minutes post-administration, subjects will be free to leave the clinic. Subjects will be instructed to keep the injection sites clean, uncovered, and to not scratch or rub the area.

In total, each subject will receive 8 intradermal injections (four per forearm), spaced two inches apart at pre-determined sites on the volar aspect of the forearms.

## 3.5. Method of Assigning Subjects to Treatment Groups

Subjects will be enrolled in parallel into 3 cohorts according to the inclusion/exclusion criteria:

- Cohort 1: 30 healthy uninfected/unexposed subjects.
- Cohort 2: 30 subjects who have recovered from SARS-CoV-2 infection at least two months prior to enrollment into the study independent of vaccination status.
- Cohort 3: 30 subjects who have received a complete SARS-CoV-2 vaccine course at least four weeks prior to enrollment into the study no known history of natural infection.

## 3.6. Blinding and Unblinding

This will be an open-label study.

#### 3.7. Schedule of Events

The full schedule of activities can be found in Table 3 of the protocol.

Version 1 

## 4. Statistical Analysis and Reporting

#### 4.1. Introduction

Data processing and tabulation of descriptive statistics will use SAS (release 9.4 or higher), unless otherwise noted. If the use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.

Continuous (quantitative) variable summaries will include the number of subjects (n) with non-missing values, mean, standard deviation (SD), median, minimum, and maximum.

Categorical (qualitative) variable summaries will include the frequency and percentage of subjects who are in the particular category or each possible value. In general, the denominator for the percentage calculation will be based upon the total number of subjects in the study population for the cohorts, or other describing characteristic, unless otherwise specified. The denominator for by-visit displays will be the number of subjects in the relevant study population with non-missing data at each visit.

The minimum and maximum will be reported with the same degree of precision (i.e., the same number of decimal places) as the observed data. Measures of location (mean and median) will be reported to 1 degree of precision more than the observed data and measures of spread (SD) will be reported to 2 degrees of precision more than the observed data.

Percentages will be presented to 1 decimal place, unless otherwise specified.

## 5. Study Halting and Stopping Rules

Dosing may be halted temporarily to investigate before the entire study is terminated. If any of the below events occur, enrollment and dosing should be paused study-wide pending review by the Sponsor, Investigator, and/or Medical Monitor. Subjects enrolled in the study must continue to be followed for the duration of the study.

- One or more subjects with a serious adverse event (SAE) considered definitely, probably, or possibly related to the IPs.
- Three or more subjects with the same or similar grade 3 or higher AEs of the same type considered definitely, probably, or possibly related to IPs.
- One AESI, considered at least possibly related to the IPs.

#### 6. Analysis Populations

The following analysis populations are planned for this study:

• **Safety Population**: includes any subjects in Cohort 1, 2, or 3 who receive at least 1 intradermal injection of the IPs. This population will be used for all safety tables.

Version 1 

- Intent-to-Treat (ITT) Population: includes any subjects in Cohort 1, 2, or 3 who provide written informed consent, satisfy all inclusion/exclusion criteria, and have a negative test result from RT-PCR detection of SARS-CoV-2 viral RNA.
- **Modified Intent-to-Treat (mITT) Population**: includes subjects from ITT who complete stages 1 and 2 of administration and have induration responses for at least one post skin test administration visit at hour 48, 72, or 96.
- Enrolled Subjects: includes subjects who have been consented and screened, with eligibility verified. This population will be used for all listings.

## 7. General Issues for Statistical Analysis

## 7.1. Statistical Definitions and Algorithms

#### 7.1.1. Baseline

The last observation recorded before the first intradermal injection of the IPs will be used as the baseline observation for all calculations of change from baseline.

## 7.1.2. Adjustments for Covariates

Not applicable to this study.

#### 7.1.3. Multiple Comparisons

There will be no adjustments for multiple comparisons.

#### 7.1.4. Handling of Dropouts or Missing Data

Any subject who withdraws from the study will not be replaced.

Unless specified otherwise in any of the previous sections, missing data will not be imputed.

#### 7.1.5. Analysis Visit Windows

Data will be summarized by nominal study visit recorded in the database.

For tabulated summaries, only the scheduled visits will be included. Unscheduled assessments will be listed.

#### 7.1.6. Derived Variables

• Change from baseline = value at current time point – value at baseline.

Version 1 

• TEAE = any adverse event with an onset date/time after the first intradermal injection of the IPs.

## 7.1.7. Data Adjustments/Handling/Conventions

Adverse events will be coded using the MedDRA version 24.0 thesaurus.

A treatment related AE is any AE with a relationship to the study drug as judged by the investigator.

#### For partial start dates:

- If the year is unknown, then do not impute the date but instead assign a missing value.
- If the year is known, but the month or month and day is unknown, then:
  - o If the year matches the year of first dose date and the end date (if present) is after first dose date, or the AE/medication is ongoing, then impute as the month and day of the first dose date. If this produces a date after the end date, assign 01 January.
  - o Otherwise, assign 01 January.
- If the year and month are known, but the day is unknown, then:
  - o If the month and year match the month and year of the first dose date, then impute as the day of the first dose date. If this produces a date after the AE/medication end date, assign 01.
  - o Otherwise, assign 01.

#### For partial end dates:

- If the year is unknown, then do not impute the date but assign as missing value.
- If the year is known but the month or month and day is unknown, then:
  - o If the year matches the year of the last date of the study (date of last contact if subject lost to follow-up; date of completion or early termination otherwise), then impute as the month and day of the last date of the study.
  - o Otherwise, assign 31 December.
- If the year and month are known, but day is unknown, then:
  - o If the month and year match the month and year of the last date of the study, then impute as the day of the last date of the study.
  - Otherwise, assign the last day of the month.

These conventions will be applied only to adverse events.

Version 1 

Missing times will be not be imputed, they will be left as missing.

## 8. Study Patients/Subjects and Demographics

### 8.1. Disposition of Patients/Subjects

Subject disposition information will be listed. Disposition for all subjects will include tabulations of the number of subjects enrolled, completing, and withdrawing, along with reasons for withdrawal, for each cohort (and overall).

#### 8.2. Protocol Violations and Deviations

Protocol deviations will be listed.

## 8.3. Demographics and Other Baseline Characteristics

Summary statistics for age, sex, ethnicity, race, height, weight, and BMI will be summarized by cohorts for subjects in the Safety population. For the continuous variables, the number of non-missing values and the mean, standard deviation, minimum, median, and maximum will be tabulated. For the categorical variables, the counts and proportions of each value will be tabulated.

Demographic and anthropometric variables (age, sex, ethnicity, race, height, weight, and BMI) will be listed by subject. In addition, medical history, smoking history, and vaccination history will be listed by subject.

## **8.4.** Exposure and Compliance

IP exposure and dosing information will be listed for each subject.

## 8.5. DTH Responses

The DTH responses will be listed for each subject by visit.

## 9. Safety Analysis

Tables for the safety analyses will be conducted on the Safety population, which includes any subjects in Cohort 1, 2, or 3 who receive at least 1 intradermal injection of the IPs. Listings will include enrolled subjects.

For this study, AESIs are anaphylactic reactions and enhanced disease from repeated exposure to SAR-CoV-2 (in subjects who have recovered from SARS-CoV-2 infection or in subjects recently vaccinated against SARS-CoV-2).

Version 1 

#### 9.1. Adverse Events

Treatment emergent AEs are defined as AEs that either commenced following initiation of study treatment or was present prior to study treatment but increased in frequency or severity following initiation of study treatment. Adverse events of special interest (AESI) include anaphylactic reaction and enhanced disease from repeated exposure to SARS-CoV-2 (in subjects who have recovered from SARS-CoV-2 infection or in subjects recently vaccinated against SARS-CoV-2).

All AEs occurring after completion of the informed consent process and before the end of study, regardless of relationship to study drug, will be included and classified by system organ class (SOC) and preferred term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA) v24.0.

For treatment-emergent AEs (TEAEs), the following will be summarized and presented for the Safety population:

An overall summary of TEAEs, which includes:

- a. the number and percentage of patients experiencing a TEAE
- b. the number and percentage of patients experiencing a TEAE by strongest relationship to IP
- c. the number and percentage of patients experiencing a TEAE by highest severity grade
- d. the number and percentage of patients experiencing a systemic allergic reaction by highest grade according to the World Allergy Organization Grading Scale for Systemic Allergy Reactions
- e. the number and percentage of patients experiencing a treatment emergent SAE (TESAE)
- f. the number and percentage of patients experiencing a TEAE leading to study discontinuation
- g. the number and percentage of patients experiencing a treatment emergent AE of Special Interest

In the overall summary of TEAEs table, besides tabulating the number and percentage of patients, the total number of TEAE episodes will also be provided. If a patient has repeated episodes of a particular TEAE, all episodes will be counted in the summary table.

All occurrences of all AEs will be listed for each patient. The listing will contain the following information: verbatim term, SOC, PT, severity (Grade1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, and Grade 4 = Potentially Life Threatening), World Allergy Organization Grading Scale for Systemic Allergic Reactions (Grades 1-5) [where applicable], relationship to study medication, date/time and day of onset, date/time and day of resolution, the outcome, whether the event was life-threatening, fatal, or a TEAE, SAE, or AESI, if it requires or prolongs hospitalization, persistent or significant disability/incapacity, congenital anomaly or birth defect,

Version 1 

or important medical event. Listings will be sorted by patient identification number, onset date, SOC, and PT. If the onset date is completely missing, these events will be presented first. If the onset date is missing a month or a day, these events will be presented before any complete dates. AEs with a relationship to study drug of possibly related will be considered related.

Local skin reaction AEs will be listed by 7-point Likert scales indicating severity of the events:

- 1 = No problem;
- 2 = Minimal problem (can be easily ignored without effort);
- 3 = Mild problem (can be ignored with effort);
- 4 = Moderate problem (cannot be ignored but does not influence my daily activities);
- 5 = Moderately severe problem (cannot be ignored and occasionally limits my daily activities);
- 6 = Severe problem (cannot be ignored and often limits my concentration on daily activities);
- 7 = Very severe problem (cannot be ignored and markedly limits my daily activities and often requires rest).

All collected data will be presented in listings.

## 9.2. Clinical Laboratory Evaluations

Individual data listings of laboratory results will be presented for each subject. Flags will be attached to the value outside of the laboratory's reference limits.

## 9.3. Vital Signs

Individual data listings of vital signs (observed and change from baseline) will be presented for each subject.

## 9.4. Physical Examination

Abnormal physical examination findings will be listed.

## 9.5. 12-Lead Electrocardiogram

12-Lead electrocardiogram interpretations will be listed.

#### 9.6. Concomitant Medication

Prior and concomitant medications will be listed. Medications that started before initial intradermal injections of investigational products will be considered prior medications whether or not they were stopped before initial intradermal injections of investigational products. Any

Version 1 

medications continuing or starting after initial intradermal injections of investigational products will be considered to be concomitant. If a medication starts before initial intradermal injections of investigational products and continues after, it will be considered both prior and concomitant.

Medications will be coded using World Organization Drug Dictionary Anatomical Therapeutic Chemical classes and preferred terms.

## 10. Changes from Planned Analysis

Because the outcome of area of induration for the DTH reactions was not as anticipated, the DTH reactions will not be statistically analyzed. Any primary, secondary, or exploratory efficacy endpoint will be omitted from the analysis and only safety will be assessed.

## 11. Other Planned Analysis

Not applicable for this study.

#### 12. References

ASA. (2018) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2018. http://www.amstat.org/about/ethicalguidelines.cfm

ICH (1998). ICH Harmonised Tripartite Guideline. Statistical Principles for Clinical Trials E9; 1998. https://database.ich.org/sites/default/files/E9\_Guideline.pdf

RSS. (2014) The Royal Statistical Society: Code of Conduct, 2014. https://rss.org.uk/about/policy-and-guidelines/code-of-conduct/.

Version 1 





#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

## **Electronic Signature Responsiblities**

You agree that your electronic signature is the equivalent of a hand-written signature and that you are responsible for actions initiated using your electronic signature. You agree to report unauthorized usage to upon discovery of such usage via email to

## Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a perpage fee. You may request delivery of such paper copies from us by following the procedure described below.

## Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

## Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to

receive required notices and consents electronically from us or to sign electronically documents from us.

## All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

| How to contact : |
|---|
| You may contact us to let us know of your changes as to how we may contact you electronically to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows: Please send an email to |
| To advise of your new email address |
| To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at and in the body of such request you must state: your previous email address, your new email address. |
| If you created a DocuSign account, you may update it with your new email address through your account preferences. |
| To request paper copies from |
| To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to and in the body of such request you must state your email address, full name, mailing address, and telephone number. |
| To withdraw your consent with |

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to and and in the body of such request you must state your email, full name, mailing address, and telephone number.

## Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

## Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by during the course of your relationship with